CLINICAL TRIAL: NCT05982379
Title: Investigation Into the Impact of Technology-Based Motivation Program Applied to the Children Followed With Cancer Diagnosis and Their Families: A Randomized Controlled Study
Brief Title: Motivation Program for Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kisecik Şengül (Other)
Responsible Party: Sponsor-Investigator, Zeynep Kisecik Şengül, Assistant Professor, Kırıkkale University
Organization: Kırıkkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ZSengul-experimental study
Record Dates: First submitted 2023-07-25; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Childhood Cancer
Keywords: Cancer; Child; Motivation; Program; Parent; Psychosocial; Technology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Among the identified strata, intervention and control groups were randomized by an independent statistician using the website www.randomizer.org. The data of the study were entered by a person other than the researcher. Statistical analysis was performed by a person other than the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This study was carried out with two groups. Technology Based Motivation Program were used for the intervention group.
  Interventions: Other: Technology Based Motivation Program
- Control (No Intervention): No application was made to the control group, standard procedure was followed.

INTERVENTIONS:
Other: Technology Based Motivation Program — A 10-week "Technology Based Motivation Program" was given to the intervention group. The website and four training modules were used with the children in the intervention group. Nine coaching interviews with each child (once a week) were conducted over WhatsApp. The children were encouraged to do progressive relaxation and breathing exercises at least twice a week, and eight therapeutic stories (once a week) were sent to the child's phone in the form of animation.
  Three training modules were used with the primary caregivers, and coaching interviews were conducted on WhatsApp twice during the program. Primary caregivers practiced progressive relaxation and breathing exercises at least twice a week. In addition, eight motivation messages were sent to the child and primary caregiver, and 24/7 consultancy was provided.
  Arms: Intervention

SUMMARY:
Purpose: To determine the effectiveness of the technology-based motivation program implemented with children with cancer diagnosis and their primary caregivers.

Methods: This randomized controlled trial was completed with 31 children and 31 primary caregivers between the ages of 9 and18, who were being treated for cancer. A 10-week "Technology Based Motivation Program" was given to the intervention group. "State/ Trait Anxiety Inventory for Children", "Paediatric Quality of Life Inventory", "Paediatric Cancer Coping Scale", "State and Trait Anxiety Inventory," and "Process Evaluation Forms" were administered. Chi-square test, Fisher-Exact test, Independent Sample-t test, Man-Whitney U test, Wilcoxon test, Pearson and Spearman correlation coefficients were used for data analysis.

DETAILED DESCRIPTION:
Design The study was conducted in two hospitals at Leukemia Polyclinic, Paediatric Haematology and Oncology Polyclinic, and Paediatric Haematology-Oncology Service from September 2019 to August 2020.

Setting and Samples In determining the research population, hospital registry information was used, and 119 children followed up with a diagnosis of cancer formed the research population. The sample of the research consisted of 44 children (leukaemia n = 33, solid tumour n = 11) and their primary caregivers meeting the inclusion criteria.

Randomization and blinding A stratified randomization method was used in the research. 44 children (leukaemia and solid tumour) who met the inclusion criteria were grouped according to gender (male and female) and age (9-13 years-14-18 years) and eight layers were obtained. Among the identified strata, intervention and control groups were randomized by an independent statistician using the website www.randomizer.org, 22 children were assigned to the intervention, and 22 to the control group. Five children from the intervention group and five children from the control group (unreachable (n=3), ex (n=1), refusal (n=4), Hematopoietic stem cell transplantation (HSCT) performed (n=1), intensive care unit admission (n=1)) could not be included in the research for various reasons and 34 children were included in the research. The purpose and content of the research were explained without informing the children and their primary caregivers that they were in the intervention or control group.

At the end of the research, the power analysis performed by using the mean scores of State Anxiety Inventory for Children with G * Power 3.0.10 program yielded a total of at least 28 samples that were found to be sufficient with 90% power and 5% margin of error (n1 = 14; n2 = 14).

Theoretical underpinnings The use of models is important in establishing the theoretical framework of research. In this research, the Transactional Stress and Coping Model of Lazarus and Folkman, which is the most widely used model in studies examining the coping and anxiety levels of children with cancer diagnosis, was used. The practices in the motivation program were created for the coping strategies of "seeking social support, self-control, positive evaluation and accepting responsibility" in the model.

Interventions The research consists of four stages. (1) Constructing training modules, (2) Creating a website, (3) Conducting preliminary intervention, and (4) Implementing the training modules with the children and primary caregivers in the intervention group.

Constructing training modules Four training modules for children and three training modules for primary caregivers were created by the researchers in line with the literature Content was added to the website after it was approved by 6 experts.

Creating the website The website was designed by a professional web design firm. The website can be accessed by computer, tablet and phone. There is an administrator and user panel on the website. Children and primary caregivers logged on the website with different passwords through the user panel and accessed the modules specially prepared for them.

Conducting preliminary intervention The preliminary intervention of the technology-based program was conducted with five children aged 9-18 years who were followed up with a diagnosis of leukaemia, and with their primary caregivers. As the child and primary caregivers found the program applicable as a result of the preliminary intervention, no change was made and it was included in the sample.

Using the training modules with children and primary caregivers in the intervention group The website and four training modules were used with the children in the intervention group. Nine coaching interviews with each child (once a week) were conducted over WhatsApp. The children were encouraged to do progressive relaxation and breathing exercises at least twice a week, and eight therapeutic stories (once a week) were sent to the child's phone in the form of animation.

Three training modules were used with the primary caregivers, and coaching interviews were conducted on WhatsApp twice during the program. Primary caregivers practiced progressive relaxation and breathing exercises at least twice a week. In addition, eight motivation messages were sent to the child and primary caregiver, and 24/7 consultancy was provided.

Control Group The routine practices of the children in the control group and their primary caregivers at the hospital continued. In addition, forms other than process evaluation were given to the child and their primary caregivers at the beginning and end of the program.

Data gathering After the children and primary caregivers who participated in the research were informed about the research in an empty room or in the room where they were treated during the polyclinic controls, data collection forms were given, the children and primary caregivers in the intervention group were subscribed to the website, and the exercises were explained in practice. It took approximately 60 minutes for the participants to fill out the forms and learn about the program. At the end of the research, the data collection forms (excluding the descriptive data form) were collected through WhatsApp messages.

Data collection tools Child and Parent Descriptive Characteristics Form, Spielberger State-Trait Anxiety Inventory, State/ Trait Anxiety Inventory for Children, Paediatric Cancer Coping Scale, Paediatric Quality of Life Inventory, and Process Evaluation Forms were used to collect the data.

Ethical considerations Permission for the research was obtained from the University Ethics Committee and Hospitals. Informed written consent was obtained from the children and their primary caregivers, who agreed to participate in the research, after written and verbal explanations were given to the patients to participate in the research. At the end of the study, all interventions were also performed with the control group.

ELIGIBILITY:
Inclusion Criteria:

For children:

* Those having received cancer treatment (leukaemia, lymphomas and solid tumours),
* Those aged 9-18 years,
* Those who speak Turkish,
* Those who have internet access on their smart phone or computer,
* Self and primary caregiver having agreed to participate in the study, and
* Those who can continue the research for 9 weeks (Trying progressive relaxation exercises, breathing exercises and imagination at least twice a week).

For primary caregivers:

* Those who speak Turkish,
* Those who are literate,
* Those who have internet access on their smart phones and computers,
* Those who agree to participate in the research, and
* Those who can continue the research for 9 weeks (Trying progressive relaxation exercises at least twice a week).

Exclusion Criteria:

* Those who do not agree to participate in the research,
* Those who have experienced significant life events in the last 6 months (migration, death, divorce etc.),
* The presence of another important disease in the family that can increase stress and prevent coping, and
* Those who do not have internet access.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Anxiety levels of the children | baseline (Initial interview) and through study completion (10th week)
  State/ Trait Anxiety Inventory for Children: 20 items for the State Anxiety, 20 items for the Trait Anxiety. The scores on the scale range from 20 to 60, and a high score indicates high anxiety.
Children's quality of life scores | baseline (Initial interview) and through study completion (10th week)
  Pediatric Quality of Life Inventory: The scale consists of 23 items and is scored from 0 to 100. The higher the score, the higher the quality of life
Coping scores of the children | baseline (Initial interview) and through study completion (10th week)
  Pediatric Cancer Coping Scale:The scale comprises 33 items related to cognitive coping, problem oriented coping, and defensive coping.The score obtained from the scale ranges from 0 to 99. Higher scores on the scale indicate a high level of coping strategies.
Anxiety levels of the primary caregivers | baseline (Initial interview) and through study completion (10th week)
  Spielberger State/ Trait Anxiety Inventory: 20 items of the 40-item scale are used to determine state anxiety and 20 items are used to determine trait anxiety.The scores on the scale range from 20 to 80, and the higher the score, the higher the level of anxiety.

SECONDARY OUTCOMES:
Application tracking forms | Every week during the intervention
  Process evaluation forms:Six forms were prepared by the researchers. It was used to follow the practices and interviews of children and primary caregivers. 1. Website training follow-up form, 2. Mobile video interview follow-up form, 3. Counseling follow-up form, 4. Children's follow-up form for interventions, 5. Primary caregivers follow-up form for interventions, 6. Satisfaction and suggestion form

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Kisecik Şengül, RN, PhD, Principal Investigator — Kırıkkale University
Locations (1):
- Zeynep Kisecik Şengül, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The confidentiality of the data used in the study will be protected.